CLINICAL TRIAL: NCT05808829
Title: The Effect of Progressive Muscle Relaxation Exercise on Mental Health and Life in University Students: A Randomized Controlled Study
Brief Title: The Effect of Progressive Relaxation Exercises in University Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Naile Bilgili, Professor, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2021-807
Record Dates: First submitted 2023-03-29; First posted 2023-04-11 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-03

CONDITIONS: Progressive Muscle Relaxation Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Research data/output measurements, analysis and reporting
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Progressive Muscle Relaxation Exercise (Experimental): Participants performed muscle relaxation exercises at least 4 times a week for 6 weeks. Once a week, the researcher exercised with the participants in online groups to control the research and to check whether the participants were doing the exercise correctly.
  Interventions: Other: Progressive Muscle Relaxation Exercise
- No Intervention: Control Group (No Intervention): The participants continued their daily life.

INTERVENTIONS:
Other: Progressive Muscle Relaxation Exercise — University students did progressive muscle relaxation exercises at least 4 times a week for 6 weeks. Once a week, exercise was done with the researcher by online interview via Zoom.
  Other Names: Progressive muscle relaxation exercise implementation, online interview
  Arms: Experimental: Progressive Muscle Relaxation Exercise

SUMMARY:
The aim of this randomized controlled study is to determine the effect of progressive muscle relaxation exercise on mental health and quality of life in university students. The research was carried out with the 1st and 2nd year students of Tokat Gaziosmanpaşa University Reşadiye Vocational School Health Care Services Department Elderly Care Program. The data of the study were collected using the Introductory Information Form, Brief Symptom Inventory, and Quality of Life Scale. University students in the intervention group were given progressive muscle relaxation exercise at least 4 times a week for 6 weeks.

DETAILED DESCRIPTION:
The aim of this randomized controlled parallel group single-center study is to determine the effect of progressive muscle relaxation exercise on mental health and quality of life in university students. The research was conducted online with Tokat Gaziosmanpaşa University Reşadiye Vocational School Health Care Services Department Aged Care Program 1st and 2nd grade students. The research was carried out with a total of 86 students, 43 of which were in the intervention group and 43 in the control group. The data of the study were collected using the Introductory Information Form, Brief Symptom Inventory, SF-36, Progressive Muscle Relaxation Exercise Follow-up Form. University students in the intervention group were given progressive muscle relaxation exercise at least 4 times a week for 6 weeks. No intervention was made in the control group. University students in the control group were asked to continue their daily lives. Ethics committee permission, institutional permission, scale usage permission and written consent of the participants were obtained for the research.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* Being 18 years or older,
* Having the necessary technology to participate in the study online (Smartphone, computer, etc.)

Exclusion Criteria:

* Presence of any diagnosed musculoskeletal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2021-08-16 (Actual); Primary Completion 2021-09-27 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Brief Symptom Inventory | 6 weeks
  Likert-type self-evaluation scale consisting of 53 items was developed to determine the mental state of individuals. Items were graded between 0-4 values corresponding to "not at all" and "too much". It consists of nine subscales, three global indexes and additional items. The 9 sub-dimensions of the scale were formed as somatization, obsessive-compulsive symptom, interpersonal sensitivity, depression, anxiety, hostility, phobic anxiety, paranoid thought and psychotism, respectively. The scale can be applied to adolescent and adult individuals and groups. The high total scores obtained from the scale indicate the frequency of the individual's symptoms. The score range is between 0-212.

SECONDARY OUTCOMES:
The Mos 36 Item Short Form Health Survey (Sf-36) | 6 weeks
  The Short Form 36 is a widely used scale in health-related quality of life research. In the evaluation of sub-dimensions; each dimension is scored between 0 and 100 points, and a high score indicates a good quality of life. The SF-36 quality of life scale consists of 8 health concepts. These are physical function, social function, role limitations due to physical problems, role limitations due to emotional problems, mental health, energy, pain and general perception of health. It consists of 36 items in total.

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University, Ankara, Çankaya/Ankara, Turkey (Türkiye)